CLINICAL TRIAL: NCT03563053
Title: Open-label, Long-term, Extension Treatment Using Intra-Erythrocyte Dexamethasone Sodium Phosphate (EryDex System) in Patients With Ataxia Telangiectasia Who Participated in the ATTeST-IEDAT-02-2015 Study
Brief Title: Extension Treatment Using EryDex System in Patients With AT Who Participated in the ATTeST-IEDAT-02-2015 Study
Acronym: OLE-IEDAT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: terminated by sponsor
Sponsor: Quince Therapeutics S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IEDAT-03-2018; 2018-000338-36 (EudraCT Number)
Record Dates: First submitted 2018-05-23; First posted 2018-06-20 (Actual); Results first posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: Ataxia Telangiectasia; Genetic Syndrome
Keywords: Ataxia Telangiectasia; AT; EryDex system; Dexamethasone; Dexamethasone sodium phosphate
MeSH Terms: conditions — Ataxia Telangiectasia; Genetic Diseases, Inborn

STUDY DESIGN:
Intervention Model Description: Open-label, Long-term, Extension Treatment
Masking Description: It's a open label extension study, so no blinding was applicable.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- active drug (Experimental): ~14-22 mg dexamethasone sodium phosphate (DSP) for 12 months. The duration of EryDex treatment could be extended further and continue until patients eventually withdrew consent, or the Investigator decided to discontinue treatment based on a risk / benefit assessment.
  Interventions: Combination Product: EryDex System

INTERVENTIONS:
Combination Product: EryDex System — EryDex System was a combination product that was used to load dexamethasone sodium phosphate (DSP) into autologous erythrocytes (EDS) creating the EDS-end product which was infused into the patients.
  EryDex treatment consisted of a dose range correspondent to the ATTeST High Dose (obtained by loading 125 mg of DSP to the EryDex process and that, in the ATTeST, resulted in a mean of 17.4 ± 5.4 mg (mean ± standard deviation) of DSP infused to patients) administered via ex vivo encapsulation into EDS that were infused into the patient with A-T.
  The dose of EryDex treatment was selected to allow collection of long-term safety data on the dose of erythrocyte encapsulated DSP that was considered more effective among the two different doses that were employed in the ATTeST study, based on the analysis of the ATTeST blinded, Phase 3 study data.

SUMMARY:
Primary Objective

To monitor and evaluate the long-term safety and tolerability of EDS-EP in AT patients.

Secondary Objective

To evaluate the long-term effect of EDS-EP on health-related Quality of Life (QoL; EQ-5D-5L scale).

Exploratory Objective:

To evaluate the long-term effect of EDS-EP in treating central nervous system (CNS) symptoms, as measured by the "Modified" International Cooperative Ataxia Rating Scale (mICARS), and Clinical Global Impression of severity and change (CGI-S/C).

DETAILED DESCRIPTION:
This was an international (North America, Europe, Africa, Asia and Australia), multi-center, prospective, open-label treatment study, designed to continue to provide the study medication to all patients who completed 12 months of treatment (including those treated with placebo) in the ATTeST-IEDAT-02-2015 trial, completed the study assessments, do not present safety contraindication to continuation of treatment, and provided informed consent.

The study aimed to collect information on the long-term safety and efficacy of the trial treatment.

Patients meeting all selection criteria received monthly infusions of EDS-EP (dose range of ~14-22 mg DSP/infusion). If this dose of EDS-EP was not tolerated, the patient was discontinued from the study.

During the study, long-term efficacy assessments were performed every 6 months, while safety parameters were assessed at each monthly visit. The Schedule of Visits and assessments for the first 12 months were replicated for the second year onwards for patients who continued EryDex treatment beyond 12 months.

The analysis of the EryDex long-term safety and tolerability was based on the occurrence of Treatment-Emergent Adverse Events (TEAEs), including Serious AEs and discontinuations due to AEs. The long-term effect was measured by the "Modified" International Cooperative Ataxia Rating Scale, (mICARS), Rescored mICARS, Clinical Global Impression of severity and change (CGI-S/C) and health-related Quality of Life (QoL; EQ-5D-5L scale).

The ICARS, EQ-5D-5L and the CGI-C / S were administered by a properly qualified rater identified at each site who performed the ratings on the efficacy measures. The ICARS rater remained blinded to other assessments and did not have access to the safety data. The CGI rater did not have access to the ICARS ratings or safety data but was able to refer to other scales in scoring the CGI.

All patients enrolled in this study have participated in Study ATTeST-IEDAT-02-2015, and there was no de novo enrollment of new patients.

EryDel S.p.A (now Quince Therapeutics) decided to discontinue the IEDAT-03-2018 study in India due to the COVID-19 pandemic. On 13 Apr 2022, after the last patient completed one year of EryDex treatment, EryDel S.p.A. communicated the end of the open label extension study IEDAT-03-2018 and the stop of the EryDex treatment for patients in the context of this study.

ELIGIBILITY:
Inclusion Criteria:

1. Patient completed the double-blind period in the ATTeST study and completed the final (Visit 15 / Month 12) Efficacy Assessments of ATTeST or discontinued the study during the COVID-19 pandemic.
2. Patient tolerated the study medication, without any evidence of steroid adverse events, or treatment-related severe events / serious adverse events.
3. Body weight > 15 kg.
4. The patient and his / her parent / caregiver (if below the age of consent), or a legal representative, provided written informed consent to participate. If consent was provided solely by the caregiver in accordance with local regulations, the patient also was asked to provide their assent to participate in the study.
5. Patient did not present safety contraindication for continuation of treatment, as determined by the Principal Investigator (PI) according to the procedures described below.

Moreover, patients who were discontinued from the ATTeST study during the COVID-19 pandemic were eligible to receive the EryDex treatment in the IEDAT-03-2018 study, in the absence of safety contraindications to continuation of the treatment, and after signing the informed consent.

There were no de novo enrolled patients.

Exclusion Criteria:

Patients who met one or more of the following criteria were not considered to be eligible to participate in the study:

General

1. Females that were:

   1. Pregnant, or were breast-feeding (for EU countries only)
   2. Of childbearing potential, pregnant, or were breast-feeding (for US and Rest of World countries).

   Females of childbearing potential using adequate birth control, as determined by their Health Care Provider, were eligible.
2. A disability that may prevent the patient from completing all study requirements.
3. Current participation in another clinical study with another investigational drug.

   Medical History and Current Status
4. Cluster differential 4 positive (CD4+) lymphocytes count < 400 / mm3 (for patients 6 years of age) or < 150 / mm3 (for patients > 6 years). In presence of oral infections, like oral candidiasis, documented at the screening or recurrent as per medical history documentation, the limit increases to < 200 / mm3 (for patients > 6 years).
5. Current neoplastic disease.
6. Severe impairment of the immunological system.
7. Severe or unstable pulmonary disease.
8. Uncontrolled diabetes. Patients with diabetes that had been stabilized (i.e., no hypoglycemic or hyperglycemic episodes in the past 3 months) were eligible.
9. Any other severe, unstable, or serious disease or condition that in the Investigator's opinion would put the patient at risk for imminent life-threatening morbidity, need for hospitalization, or mortality.
10. Eligibility of patients with abnormal laboratory test values were determined by the Investigator.
11. Confirmed haemoglobinopathies, e.g., haemoglobin C disease, sickle cell anaemia, or thalassemia.
12. Moderate or severe renal and / or hepatic impairment.
13. Patients who experienced moderate / severe steroid side effects, or moderate / severe adverse events associated with the EryDex treatment administered in the ATTeST study.

    Prior / Concomitant Medication
14. Requires treatment with an oral or parenteral steroid. Treatment with inhaled or intranasal steroids for asthma or allergies, as well as use of topical steroids were permitted.
15. Requires any other concomitant medication prohibited by the protocol.
16. Use of any drug that is a strong inducer / inhibitor of Cytochrome P450 3A4 (CYP3A4).

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2022-09-02 (Actual); Study Completion 2022-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guenter R Janhofer, MD, PhD, Study Director — EryDel S.p.A.
Locations (17):
- United States (4):
  - Ataxia Center and HD Center of Excellence - UCLA, Los Angeles, California
  - Division of Pediatric Allergy and Immunology - Johns Hopkins Hospital, Baltimore, Maryland
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Department of Pediatrics Division of Child and Adolescent Neurology Mitochondrial Clinic - University of Texas Medical School, Houston, Texas
- Department of Neurology Royal Children's Hospital, Parkville, Victoria, Australia
- Laboratory of Pediatric Immunology UZ Leuven, Leuven, Belgium
- Klinik für Kinder- und Jugendmedizin, Allergologie, pneumologie und Mukoviszidose, Universitätsklinikum Frankfurt, Frankfurt, Germany
- India (4):
  - Vijaya Health Centre, Department of Neurology, Chennai, Tamil Nadu
  - National Institute of Mental Health and Neurosciences (NIMHANS) Department of Neurology, Bangalore
  - Nizam's Institute of Medical Sciences Department of Neurology, Hyderabad
  - Jaslok Hospital and Research Center Department of Pediatric Neurology, Mumbai
- Dipartimento Neuroscienze umane e salute mentale, Policlinico Umberto I Università La Sapienza, Roma, Italy
- Norwegian National Unit for Newborn Screening, Division of Pediatric and Adolescent Medicine, Oslo University Hospital, Oslo, Norway
- Department of Clinical Immunology - The Children's Memorial Health Institute, Warsaw, Poland
- Servicio de Neurolgia Pediatrica, Hospital Materno-Infantil La Paz, Madrid, Spain
- Razi Hospital, Clinical Investigation Center-Neuroscience, Tunis, Tunisia
- Nottingham University Hospitals NHS Trust - Queen's Medical Centre, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Koenig MK, Leuzzi V, Gouider R, Yiu EM, Pietrucha B, Stray-Pedersen A, Perlman SL, Wu S, Burgers T, Borgohain R, Kandadai RM, Meyts I, Bucciol G, Udwadia-Hegde A, Yadav R, Roberts D, Dane A, Roden M, Thye D, Horn B, Lederman HM, Whitehouse WP. Long-term safety of dexamethasone sodium phosphate encapsulated in autologous erythrocytes in pediatric patients with ataxia telangiectasia. Front Neurol. 2025 Jan 23;15:1526914. doi: 10.3389/fneur.2024.1526914. eCollection 2024. PMID 39917433

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Out of a total of 108 patients who completed the full treatment period (including placebo treatment) in the ATTeST - IEDAT-02 study, 104 patients were enrolled in the IEDAT-03-2018 study (OLE-IEDAT) and comprised the Total Set. These patients signed the ICF, completed the ATTeST study assessments, and did not present safety contraindication prior continuation with the EryDex treatment.
Groups:
- Active Drug: ~14-22 mg dexamethasone sodium phosphate (DSP) for 12 months. The duration of EryDex treatment could be extended further and continue until patients eventually withdrew consent, or the Investigator decided to discontinue treatment based on a risk / benefit assessment.
  EryDex System: EryDex System is a combination product that is used to load dexamethasone sodium phosphate (DSP) into autologous erythrocytes (EDS) creating the EDS-end product which is infused into the patients.
  EryDex treatment consisted of a dose range correspondent to the ATTeST High Dose (obtained by loading 125 mg of DSP to the EryDex process and that, in the ATTeST, resulted in a mean of 17.4 ± 5.4 mg (mean ± standard deviation) of DSP infused to patients) administered via ex vivo encapsulation into EDS that were infused into the patient with A-T. The dose of EryDex treatment was selected to allow collection of long-term safety data on the dose of erythrocyte encapsulated DSP that was considered more effective among the two different doses that were employed in the ATTeST study, based on the analysis of the ATTeST blinded, Phase 3 study data.
Period: Overall Study
Arm/Group | Active Drug
Started | 104
Total Set | 104
Safety Set | 104
Full Analysis Set | 80
Month 12 | 64
Month 24 | 33
Month 36 | 21
Month 48 | 7
Month 50.5 | 1
Completed | 0
Not Completed | 104
Not completed — Withdrawal by Subject | 17
Not completed — Due to the COVID-19 pandemic | 12
Not completed — Adverse Event | 3
Not completed — Physician Decision | 1
Not completed — study terminated by sponsor | 71

BASELINE CHARACTERISTICS:
Population: In this trial, the Total or Overall Set (N=104) numerically corresponds to the Safety set, which included all patients who provided informed consent or assent and who received any dose of study medication during ATTeST-IEDAT-03-2018 study (i.e., "Date performed" given on the "EDS-EP Infusion" eCRF page at any Visit).
Groups:
- Overall Population (Total Set): The Total Set (N=104) included all patients who provided informed consent or assent as documented by a date of informed consent or date of assent on the 'Informed Consent' Electronic Case Report form (eCRF) page.
Arm/Group | Overall Population (Total Set)
Number analyzed (Participants) | 104
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 104
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.4 (4.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 55
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 99
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 21
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 80
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Belgium | 3
  United States | 25
  Poland | 10
  Italy | 2
  Australia | 2
  Tunisia | 7
  Germany | 13
  India | 15
  Spain | 11
  Norway | 5
  United Kingdom | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment-Emergent Adverse Event (TEAE), Treatment-emergent Serious Adverse Events (TESAE), and Adverse Events of Special Interest (AESI) Throughout the Study
Description: Assessment of TEAEs, treatment-emergent serious adverse events (TESAE), and adverse events of special interest (AESI) were performed throughout the study, from the time of signing of the ICF at Baseline Visit through to the Final Study Visit (Month 12 or early discontinuation). All patients were to be followed up through 30 days after the Final Visit (Month 12 or early discontinuation) or at least 60 days after the final infusion, whichever was longer.
Time Frame: From Baseline (Visit 1 - Day 0) to Follow-up (~60 days after last infusion, i.e. up to 50.5 months)
Population: Safety Population (SAF): the Safety Analysis Set consisted of all patients who provided informed consent or assent and who received any dose of study medication during IEDAT-03-2018 study. The Safety Analysis Set was used for all safety analyses.
Measure: Number; unit: Number of events
Groups:
- Overall Population (SAF): The Total Set (N=104) included all patients who provided informed consent or assent as documented by a date of informed consent or date of assent on the 'Informed Consent' Electronic Case Report form (eCRF) page.
Arm/Group | Overall Population (SAF)
Number analyzed (Participants) | 104
Number of events
  Number of TEAEs | 1232
  Number of Serious TEAEs | 19
  Number of TEAE leading to Death | 0
  Number of TEAE leading to Permanent Withdrawal of Treatment | 5
  Adverse Events During COVID-19 Interruption - On Dose | 5
  Adverse Events During COVID-19 Interruption - Off Dose | 3
  Adverse Events During COVID-19 Interruption - Restart | 55
  TEAE by Worst Intensity - Mild | 1028
  TEAE by Worst Intensity - Moderate | 187
  TEAE by Worst Intensity - Severe | 17
  TEAE by Closest Relationship to Treatment - Probable | 283
  TEAE by Closest Relationship to Treatment - Possible | 167
  TEAE by Closest Relationship to Treatment - Unlikely | 178
  TEAE by Closest Relationship to Treatment - Not related | 604
  Number of AESI | 83

2. Secondary Outcome: Change From Baseline in Quality of Life Using EQ-5D-5L Scale to Month 36
Description: The EQ-5D included single item measures of 5 health dimensions:
  * mobility,
  * self-care,
  * usual activities,
  * pain / discomfort, and
  * anxiety / depression. The EQ-5D-5L included five levels of severity (i.e., no problems, slight problems, moderate problems, severe problems, and extreme problems) for each of the five EQ-5D dimensions. These levels were scored from 1 = no problems to 5 = extreme problems: from 5, min/worst, to 25, best/max).The EQ-5D results were converted into a continuous index score: as for this index score, the closer the value is to 1, the better is the health status.
  The efficacy data focus mainly up to Month 36 as afterwards the number of patients / assessments dropped below 20% of the initial sample size, which was required for the efficacy evaluations.
Time Frame: From Baseline (Visit 1- Day 0) to Month 36
Population: Full Analysis Set Population (FAS): the FAS comprised all patients who entered IEDAT-03-2018 study, had a Baseline Efficacy Assessment in IEDAT-03-2018 and who received at least one dose of study medication and had at least one post-Baseline Efficacy Assessment of the ICARS in this extension study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Overall Population (Total Set)
Number analyzed (Participants) | 80
score on a scale
  to Month 6: number analyzed (Participants) | 73
  to Month 6 | 0.015 (0.1131)
  to Month 12: number analyzed (Participants) | 61
  to Month 12 | -0.022 (0.1145)
  to Month 18: number analyzed (Participants) | 51
  to Month 18 | 0.007 (0.1233)
  to Month 24: number analyzed (Participants) | 32
  to Month 24 | 0.011 (0.1746)
  to Month 30: number analyzed (Participants) | 22
  to Month 30 | -0.021 (0.1117)
  to Month 36: number analyzed (Participants) | 20
  to Month 36 | 0.011 (0.1242)

3. Secondary Outcome: Number of Patients With Improving, Stable or Worsening Score Using a Clinical Global Impression of Change (CGI-C) From Baseline (Visit 1- Day 0) to Month 36
Description: The CGI-C scale assesses the change in the patient's clinical status from baseline using a 7-point scale, ranging from 1 (very much improved) to 7 (very much worse), with a score of 4 indicating no change. Clinicians were required to conduct a full clinical interview and examination of the patient.
  The interview and examination assessed various aspects of the patient's appearance (grooming, evidence of falls, etc.), ataxia, cognition (orientation, calculation ability, language, ability to follow commands, memory, etc.), apraxia, dysarthria, extrapyramidal motor symptoms, activities of daily living, and mood. The higher the score the worse the outcome.
  The efficacy data focus mainly up to Month 36 as afterwards the number of patients / assessments dropped below 20% of the initial sample size, which was required for the efficacy evaluations.
Time Frame: From Baseline (Visit 1- Day 0) to Month 36
Population: The FAS comprised all patients who entered IEDAT-03-2018 study, had a Baseline Efficacy Assessment in IEDAT-03-2018 and who received at least one dose of study medication and had at least one post-Baseline Efficacy Assessment of the ICARS in this extension study.
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Population (Total Set)
Number analyzed (Participants) | 80
Participants
  Month 6 - Improved (Score 1-3): number analyzed (Participants) | 77
  Month 6 - Improved (Score 1-3) | 9
  Month 6 - No change or Worsened (Score 4-7): number analyzed (Participants) | 77
  Month 6 - No change or Worsened (Score 4-7) | 68
  Month 12 - Improved (Score 1-3): number analyzed (Participants) | 59
  Month 12 - Improved (Score 1-3) | 14
  Month 12 - No change or Worsened (Score 4-7): number analyzed (Participants) | 59
  Month 12 - No change or Worsened (Score 4-7) | 45
  Month 18 - Improved (Score 1-3): number analyzed (Participants) | 47
  Month 18 - Improved (Score 1-3) | 6
  Month 18 - No change or Worsened (Score 4-7): number analyzed (Participants) | 47
  Month 18 - No change or Worsened (Score 4-7) | 41
  Month 24 - Improved (Score 1-3): number analyzed (Participants) | 31
  Month 24 - Improved (Score 1-3) | 5
  Month 24 - No change or Worsened (Score 4-7): number analyzed (Participants) | 31
  Month 24 - No change or Worsened (Score 4-7) | 26
  Month 30 - Improved (Score 1-3): number analyzed (Participants) | 19
  Month 30 - Improved (Score 1-3) | 2
  Month 30 - No change or Worsened (Score 4-7): number analyzed (Participants) | 19
  Month 30 - No change or Worsened (Score 4-7) | 17
  Month 36 - Improved (Score 1-3): number analyzed (Participants) | 19
  Month 36 - Improved (Score 1-3) | 3
  Month 36 - No change or Worsened (Score 4-7): number analyzed (Participants) | 19
  Month 36 - No change or Worsened (Score 4-7) | 16

4. Secondary Outcome: Number of Patients With None to Severe (0 to 4) Scores in Clinical Global Impression of Severity (CGI-S)-Structured of Neurological Symptoms of AT From Baseline (Visit 1 - Day 0) to Month 36
Description: The CGI-S scale measures global severity of illness at a given point in time, and is usually rated on a 7-point, Likert-type scale ranging from 1 (normal, not ill at all) to 7 (among the most extremely ill patients). No version of the CGI-S exists which has been specifically adapted for use in patients with A-T; therefore, a 5-point version was developed that considered the severity of the following symptoms of A-T: ataxia (walking), dysarthria, dysmetria, extrapyramidal symptoms (chorea, myoclonus, dystonia, and tremor), and eye movements. Ratings of none (0), mild (1), moderate (2), severe (3), and very severe (4) were selected based on the level of symptomatology. The higher the score the worse the outcome.
  The efficacy data focus mainly up to Month 36 as afterwards the number of patients / assessments dropped below 20% of the initial sample size, which was required for the efficacy evaluations.
Time Frame: From Baseline (Visit 1- Day 0) to Month 36
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Population (Total Set)
Number analyzed (Participants) | 80
Participants
  Baseline - CGI-S Score - 0: number analyzed (Participants) | 74
  Baseline - CGI-S Score - 0 | 2
  Baseline - CGI-S Score - 1: number analyzed (Participants) | 74
  Baseline - CGI-S Score - 1 | 18
  Baseline - CGI-S Score - 2: number analyzed (Participants) | 74
  Baseline - CGI-S Score - 2 | 31
  Baseline - CGI-S Score - 3: number analyzed (Participants) | 74
  Baseline - CGI-S Score - 3 | 23
  Baseline - CGI-S Score - 4: number analyzed (Participants) | 74
  Baseline - CGI-S Score - 4 | 0
  Month 6 - CGI-S Score - 0: number analyzed (Participants) | 76
  Month 6 - CGI-S Score - 0 | 1
  Month 6 - CGI-S Score - 1: number analyzed (Participants) | 76
  Month 6 - CGI-S Score - 1 | 20
  Month 6 - CGI-S Score - 2: number analyzed (Participants) | 76
  Month 6 - CGI-S Score - 2 | 30
  Month 6 - CGI-S Score - 3: number analyzed (Participants) | 76
  Month 6 - CGI-S Score - 3 | 22
  Month 6 - CGI-S Score - 4: number analyzed (Participants) | 76
  Month 6 - CGI-S Score - 4 | 3
  Month 12 - CGI-S Score - 0: number analyzed (Participants) | 59
  Month 12 - CGI-S Score - 0 | 0
  Month 12 - CGI-S Score - 1: number analyzed (Participants) | 59
  Month 12 - CGI-S Score - 1 | 12
  Month 12 - CGI-S Score - 2: number analyzed (Participants) | 59
  Month 12 - CGI-S Score - 2 | 28
  Month 12 - CGI-S Score - 3: number analyzed (Participants) | 59
  Month 12 - CGI-S Score - 3 | 17
  Month 12 - CGI-S Score - 4: number analyzed (Participants) | 59
  Month 12 - CGI-S Score - 4 | 2
  Month 18 - CGI-S Score - 0: number analyzed (Participants) | 47
  Month 18 - CGI-S Score - 0 | 0
  Month 18 - CGI-S Score - 1: number analyzed (Participants) | 47
  Month 18 - CGI-S Score - 1 | 13
  Month 18 - CGI-S Score - 2: number analyzed (Participants) | 47
  Month 18 - CGI-S Score - 2 | 21
  Month 18 - CGI-S Score - 3: number analyzed (Participants) | 47
  Month 18 - CGI-S Score - 3 | 12
  Month 18 - CGI-S Score - 4: number analyzed (Participants) | 47
  Month 18 - CGI-S Score - 4 | 1
  Month 24 - CGI-S Score - 0: number analyzed (Participants) | 31
  Month 24 - CGI-S Score - 0 | 0
  Month 24 - CGI-S Score - 1: number analyzed (Participants) | 31
  Month 24 - CGI-S Score - 1 | 10
  Month 24 - CGI-S Score - 2: number analyzed (Participants) | 31
  Month 24 - CGI-S Score - 2 | 10
  Month 24 - CGI-S Score - 3: number analyzed (Participants) | 31
  Month 24 - CGI-S Score - 3 | 9
  Month 24 - CGI-S Score - 4: number analyzed (Participants) | 31
  Month 24 - CGI-S Score - 4 | 2
  Month 30 - CGI-S Score - 0: number analyzed (Participants) | 19
  Month 30 - CGI-S Score - 0 | 0
  Month 30 - CGI-S Score - 1: number analyzed (Participants) | 19
  Month 30 - CGI-S Score - 1 | 5
  Month 30 - CGI-S Score - 2: number analyzed (Participants) | 19
  Month 30 - CGI-S Score - 2 | 10
  Month 30 - CGI-S Score - 3: number analyzed (Participants) | 19
  Month 30 - CGI-S Score - 3 | 4
  Month 30 - CGI-S Score - 4: number analyzed (Participants) | 19
  Month 30 - CGI-S Score - 4 | 0
  Month 36 - CGI-S Score - 0: number analyzed (Participants) | 19
  Month 36 - CGI-S Score - 0 | 0
  Month 36 - CGI-S Score - 1: number analyzed (Participants) | 19
  Month 36 - CGI-S Score - 1 | 3
  Month 36 - CGI-S Score - 2: number analyzed (Participants) | 19
  Month 36 - CGI-S Score - 2 | 10
  Month 36 - CGI-S Score - 3: number analyzed (Participants) | 19
  Month 36 - CGI-S Score - 3 | 6
  Month 36 - CGI-S Score - 4: number analyzed (Participants) | 19
  Month 36 - CGI-S Score - 4 | 0

5. Secondary Outcome: Change From Baseline of the Modified International Cooperative Ataxia Rating Scale (mICARS) Until Month 36
Description: The International Cooperative Ataxia Rating Scale (ICARS) was an assessment of the degree of impairment in patients with cerebellar ataxia and was administered in its entirety; however, the primary efficacy assessment was based on the modified (m)ICARS, which excluded the Oculomotor domain (items 17 to 19) and items 8 to 12 of the Kinetic Functions domain of the ICARS. The mICARS was a 54 points maximum score (min 0) questionnaire divided into 3 sections:
  * Posture and Gait Disturbance section-7 items (min score 0, max score 34)
  * Kinetic Function-2 items (min 0, max 12)
  * Speech Disorder- 2 items (min 0, max 8). An higher scores - both for total and subscores - indicate a higher level of disease impairment. The subscores are added to give the total score.
  The efficacy data focus mainly up to Month 36 as afterwards the number of patients / assessments dropped below 20% of the initial sample size, which was required for the efficacy evaluations.
Time Frame: From Baseline (Visit 1- Day 0) to Month 36
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Overall Population (Total Set)
Number analyzed (Participants) | 80
score on a scale
  to Month 6: number analyzed (Participants) | 78
  to Month 6 | 0.7 (4.09)
  to Month 12: number analyzed (Participants) | 60
  to Month 12 | 1.5 (3.36)
  to Month 18: number analyzed (Participants) | 48
  to Month 18 | 2.7 (4.28)
  to Month 24: number analyzed (Participants) | 32
  to Month 24 | 3.9 (4.96)
  to Month 30: number analyzed (Participants) | 21
  to Month 30 | 4.5 (5.41)
  to Month 36: number analyzed (Participants) | 18
  to Month 36 | 34.0 (5.17)

ADVERSE EVENTS:
Time Frame: TEAEs were all the AEs reported from Baseline (Visit 1 - Day 0) to Follow-up (~60 days after last infusion, i.e. up to 50.5 months).
Description: All AEs that occurred during this IEDAT-03-2018 study are defined as TEAEs, as all patients received EryDex treatment in the study.
Groups:
- Overall Population (SAF): The Safety Analysis Set consisted of all patients who provided informed consent or assent and who received any dose of study medication during IEDAT-03-2018 study . The Safety Analysis Set was used for all safety analyses.
Arm/Group | Overall Population (SAF)
All-Cause Mortality (participants affected / at risk) | 0/104
Serious Adverse Events (participants affected / at risk) | 12/104
Other Adverse Events (participants affected / at risk) | 98/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Population (SAF) (N=104)
Lower respiratory tract infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
B-Cell limphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hodgkin's Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Odontogenic cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 2 (2)
Trombocytopenic Purpura (Blood and lymphatic system disorders) | 1 (5)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 1 (2)
Central nervous system lesion (Nervous system disorders) | 1 (1)
Pharyngeal swelling (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Gastrointestinal Tube Insertion (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Population (SAF) (N=104)
Upper respiratory tract infection (Infections and infestations) | 23 (36)
Nasopharyngitis (Infections and infestations) | 21 (30)
Corona Virus Infection (Infections and infestations) | 17 (19)
Bronchitis (Infections and infestations) | 10 (15)
Urinary Tract Infection (Infections and infestations) | 6 (7)
Pyrexia (General disorders) | 33 (54)
Fatigue (General disorders) | 16 (20)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 28 (199)
Fall (Injury, poisoning and procedural complications) | 7 (10)
Diarrhoea (Gastrointestinal disorders) | 23 (32)
Vomiting (Gastrointestinal disorders) | 20 (38)
Nausea (Gastrointestinal disorders) | 7 (9)
Rash (Skin and subcutaneous tissue disorders) | 9 (11)
Erythema (Skin and subcutaneous tissue disorders) | 7 (10)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 19 (42)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 12 (17)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 (10)
Serum Ferritin Decreased (Investigations) | 8 (9)
Coronavirus Test Positive (Investigations) | 7 (8)
Blood Lactate Dehydrogenase Increased (Investigations) | 6 (8)
Headache (Nervous system disorders) | 15 (22)
Iron Deficiency (Metabolism and nutrition disorders) | 16 (29)
Anaemia (Blood and lymphatic system disorders) | 6 (9)
Product contamination (Product Issues) | 13 (19)
Skin Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (10)

LIMITATIONS AND CAVEATS:
India was particularly affected by COVID-19-dependent treatment and visit interruptions.This long interruption would have resulted in insufficient long-term safety data. For this reason, EryDel (now Quince Therapeutics) decided to discontinue the IEDAT-03-2018 study in India.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-12-01): https://cdn.clinicaltrials.gov/large-docs/53/NCT03563053/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-25): https://cdn.clinicaltrials.gov/large-docs/53/NCT03563053/SAP_001.pdf